CLINICAL TRIAL: NCT04026763
Title: MR/TRUS Fusion Guided Prostate Biopsy- An Improved Way To Detect And Quantify Prostate Cancer
Brief Title: MR/TRUS Fusion Guided Prostate Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Ardeshir R Rastinehad, Associate Professor of Radiology and Urology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 15-0768
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Prostate Disease; Elevated Prostate Specific Antigen; Family History of Prostate Cancer; Positive Digital Rectal Exam
Keywords: Targeted Prostate Biopsy
MeSH Terms: conditions — Prostatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Males with Prostate Cancer (Experimental): Each participant will receive standard of care prostate biopsy as well as a US guided prostate biopsy and a MR/TRUS Fusion Guided prostate biopsy guided prostate biopsy.
  Interventions: Procedure: prostate biopsy; Procedure: MR US Fusion Guided Prostate Biopsy; Device: MR/TRUS Fusion Guided Prostate Biopsy

INTERVENTIONS:
Procedure: prostate biopsy — standard of care
Procedure: MR US Fusion Guided Prostate Biopsy — Trans-rectal ultrasound (TRUS) guided fusion prostate biopsy, Transperineal Ultrasound guided fusion prostate biopsy
  Other Names: Fusion Biopsy
Device: MR/TRUS Fusion Guided Prostate Biopsy — TRUS images are overlaid on a previously obtained prostate MRI, combined with an electromagnetic tracking system. The urologist then performs directed prostate biopsies at MR-identified targets in addition to the standard prostate biopsies.

SUMMARY:
This study will determine if targeted (Magnetic Resonance (MR) / Ultrasound (US) fusion biopsy) plus conventional biopsy is superior to conventional biopsy alone in diagnosing subjects with prostate cancer.

DETAILED DESCRIPTION:
The efficacy of targeting lesions for surgery may be limited by the visibility of a target during the procedure. The successful outcome of surgical intervention depends upon accurate device placement, which may be very challenging in certain settings, such as when a kidney tumor only is visible for a brief moment during the transient arterial phase of a contrast injection, and soon disappearing on dynamic imaging.

Historically, prostate cancer was diagnosed by digitally guided trans-rectal prostate biopsies. With PSA (Prostate Specific Antigen) screening and improvements in ultrasonography, trans-rectal ultrasound (TRUS) guided prostate biopsy have become the standard of care to screen and diagnose localized prostate cancer. Standard US 12-14 core prostate biopsy is now common practice, detecting cancer in 27% to 44% of patients.

Prostate MR imaging at 3 Tesla magnet dramatically improves diagnostic utility dramatically but biopsies are difficult, time-consuming, and require specialized equipment, which increases the cost significantly.

To meet this challenge TRUS images are overlaid on a previously obtained prostate MRI, combined with an electromagnetic tracking system. The urologist then performs directed prostate biopsies at MR-identified targets in addition to the standard prostate biopsies.

This study will consist of comparison of the standard of care prostate biopsy with the protocol biopsy which consists of a US guided prostate biopsy and a MR/US fusion tracked prostate biopsy. Each patient will act as their own control.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a pre-operative MRI performed in accordance with the MT Sinai/NIH MR prostate imaging guidelines.
* Age greater than 18 years.
* No serious concurrent medical illness that would preclude the patient from making a rational informed decision on participation.
* The ability to understand and willingness to sign a written informed consent form, and to comply with the protocol. If in question, an ethics consult will be obtained.
* Ability to tolerate sedation and or general anesthesia if required.
* PSA >2.5 or Abnormal digital rectal exam or current recommendations for biopsy from the American Urological Association
* Pre-biopsy prostate MRI as described above, showing targetable lesions within 4 months of biopsy
* Able to tolerate a ultrasound guided biopsy

Exclusion Criteria:

* Patients with an altered mental status that precludes understanding or consenting for the biopsy procedure will be excluded from this study.
* Patients unlikely able to hold reasonably still on a procedure table for the length of the procedure.
* Patients with pacemakers or automatic implantable cardiac defibrillators (contraindications to MRI)
* Patients with uncorrectable coagulopathies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Prostate Cancer | Day 0 - day of procedure
  Incidence of diagnosing subjects with prostate cancer with MR visible lesions

SECONDARY OUTCOMES:
Incidence of adverse events | 1 month
  the incidence of adverse events occurring after a targeted and ultrasound guided prostate biopsy
Pirads score | 1 month
  The Prostate Imaging Reporting and Data System (PIRADS) score classifies MRI lesions on a scale from 1 to 5, which reflects their level of suspicion from least to most. Higher score indicates more suspicion.
Gleason score | 1 month
  The Gleason Score ranges from 1-5 and describes how much the cancer from a biopsy looks like healthy tissue (lower score) or abnormal tissue (higher score). Sum of the gleason grade of the most predominant tumor pattern and a second gleason grade of the second most predominant pattern. Full score from 2 to 10, with higher score indicating more clinically significance.

CONTACTS AND LOCATIONS:
Overall Officials: Ardeshir Rastinehad, DO, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Winoker JS, Wajswol E, Falagario U, Maritini A, Moshier E, Voutsinas N, Knauer CJ, Sfakianos JP, Lewis SC, Taouli BA, Rastinehad AR. Transperineal Versus Transrectal Targeted Biopsy With Use of Electromagnetically-tracked MR/US Fusion Guidance Platform for the Detection of Clinically Significant Prostate Cancer. Urology. 2020 Dec;146:278-286. doi: 10.1016/j.urology.2020.07.072. Epub 2020 Sep 18. PMID 32956688